CLINICAL TRIAL: NCT01527461
Title: Identifying Unique Scent Signature of Lung Cancer Through Body Odor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Nir Peled MD, PhD, Head, Thoracic Cancer Research and Detection Center,Tel Hashomer, Israel, Sheba Medical Center
Other Study IDs: SHEBA-11-9031-NP-CTIL
Record Dates: First submitted 2012-01-27; First posted 2012-02-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Lung Neoplasms
Keywords: lung neoplasms; dogs; sweat; smell
MeSH Terms: conditions — Lung Neoplasms; Anosmia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sweat samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer Patients: diagnosed lung cancer patients .
- COPD Patients: COPD patients, not diagnosed with lung cancer.

SUMMARY:
The purpose of this study is to show that dogs are able to detect cancer in sweat samples. This potentially would be the base for developing a new efficient, non invasive and inexpensive diagnosis tool of lung cancer.

DETAILED DESCRIPTION:
Among all cancers which harm the population, lung cancer is the most lethal type, responsible for 1.3 million deaths per year worldwide, for 28% of all cancer deaths.The 5 year survival rates are low, only 15%.

Diagnosis and treatment of lung cancer in its early stages could increase the 5-year-survival rate by 3-4 fold with a potential for cure. Therefore, efforts are being made to develop new sensitive specified screening tools for detecting lung cancer at its' earliest stages.

A new emerging strategy for early detection of lung cancer is based on the recognition of the tumors metabolic signature, on the identification of specific biomarkers for the disease, such as the volatile organic compounds (VOC). Research has demonstrated that these compounds are released from the cancerous tissue from the early stages of the disease, and can be found in different bodily secretions.

The subjects, lung cancer patients and chronic obstructive pulmonary disease (COPD) patients, would be given cotton T-shirts with instructions to wear them without previously applying deodorant or any other similar personal hygiene products. Then, the shirts would be collected and 8 pieces (size:1cm*3cm from the armpit areas) would be cut from each one.

Dogs for this study would be trained by the "Dogs for People" association. In the initial stage, 40 mixed breed dogs and 3-4 Springer spaniels would be exposed to sweat sample collected from cancer patients in order to get them acquainted with the scent. Then, it would be demanded of them to locate boxes containing T-shirt sample taken from cancer patients, from decoy boxes holding naïve T-shirts. Every sequence will include 4 boxes with a different ratio between the specimens(each time a different number of boxes will contain samples taken from cancer patients, 0,1,2,3 or 4 when the rest of the boxes would contain naïve T-shirts). The dogs would mark the specimen by sitting next to each relevant box (they will ignore the decoy boxes after sniffing them and identifying them as irrelevant).

The most prominent 8-9 dogs would continue to the experiment phase. Each training course would last for 5-10 minutes or for 8 successful identifications, depending on the training dog needs. Dogs would be rewarded with a treat (a dog biscuit) or with play time, depending on the dogs' nature.

In the experimental phase, the decoy boxes would hold sweat samples collected from COPD patients instead of naïve T-shirts. The dogs would be asked to locate boxes containing the T-shirt sample taken from the lung cancer patients, from the decoy boxes. Every sequence will include 4 boxes with a different ratio between the specimens (each time a different number of boxes will contain samples taken from cancer patients, 0,1,2,3 or 4 when the rest of the boxes would contain samples collected from COPD patients). The dogs would mark the specimen by sitting next to each relevant box (they will ignore the decoy boxes after sniffing them and identifying them as irrelevant).

The trainer would be oblivious to the targets' location.

ELIGIBILITY:
Inclusion Criteria:

• A diagnosis of lung cancer, regardless of histology.

Exclusion Criteria

* Inability to comply with study and/or follow up procedure.
* Co morbidity of lung cancer and an additional malignancy combined.
* Patients taking part in another clinical trial and receiving any treatment for it.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The recruitment process will take place at the lung department of Sheba medical center. The participating physicians will enroll the patients and sing them on the consent form when they come for their regular appointments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02

PRIMARY OUTCOMES:
Number of patients with lung neoplasms | one year
  Dogs ability to distinguish between COPD and lung cancer patients sweat samples

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Hasomer, Israel